CLINICAL TRIAL: NCT05998798
Title: A Journey Endometrial Cancer Clinical Trials - Revealing Engagement Patterns Among Individuals Affected by Endometrial Cancer
Brief Title: Revealing Engagement Patterns Among Endometrial Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82379206
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study intends to investigate the personal experiences of endometrial cancer patients who take part in a separate clinical study including a specific medication intervention. The major focus will be on closely following individuals' rates of trial completion and withdrawal.

The data collected from this study will help improve future outcomes for all endometrial cancer patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with endometrial cancer
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endometrial cancer who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an endometrial cancer clinical research | 3 months
Rate of patients who remain in an endometrial cancer clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Malley DM, Bariani GM, Cassier PA, Marabelle A, Hansen AR, De Jesus Acosta A, Miller WH Jr, Safra T, Italiano A, Mileshkin L, Xu L, Jin F, Norwood K, Maio M. Pembrolizumab in Patients With Microsatellite Instability-High Advanced Endometrial Cancer: Results From the KEYNOTE-158 Study. J Clin Oncol. 2022 Mar 1;40(7):752-761. doi: 10.1200/JCO.21.01874. Epub 2022 Jan 6. PMID 34990208
- [Background] Marth C, Tarnawski R, Tyulyandina A, Pignata S, Gilbert L, Kaen D, Rubio MJ, Frentzas S, Beiner M, Magallanes-Maciel M, Farrelly L, Choi CH, Berger R, Lee C, Vulsteke C, Hasegawa K, Braicu EI, Wu X, McKenzie J, Lee JJ, Makker V. Phase 3, randomized, open-label study of pembrolizumab plus lenvatinib versus chemotherapy for first-line treatment of advanced or recurrent endometrial cancer: ENGOT-en9/LEAP-001. Int J Gynecol Cancer. 2022 Jan;32(1):93-100. doi: 10.1136/ijgc-2021-003017. Epub 2021 Nov 19. PMID 34799418
- [Background] Stelloo E, Nout RA, Osse EM, Jurgenliemk-Schulz IJ, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Nijman HW, Putter H, Bosse T, Creutzberg CL, Smit VT. Improved Risk Assessment by Integrating Molecular and Clinicopathological Factors in Early-stage Endometrial Cancer-Combined Analysis of the PORTEC Cohorts. Clin Cancer Res. 2016 Aug 15;22(16):4215-24. doi: 10.1158/1078-0432.CCR-15-2878. Epub 2016 Mar 22. PMID 27006490

DOCUMENTS (1):
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT05998798/ICF_000.pdf